CLINICAL TRIAL: NCT06099002
Title: Balance, Walking Speed, Quadriceps Femoris Muscle Strength and Quality of Life in Falling and Non-falling Individuals With COPD
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meral SERTEL, associate professor, Kırıkkale University
Other Study IDs: KKU-FTR-YK-02
Record Dates: First submitted 2023-09-12; First posted 2023-10-25 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with COPD over the age of 65 with a history of falls: Individuals with COPD who were over the age of 65 and had a history of falling were included in this group.
  Interventions: Other: Changed Medical research Council,Mini Mental Test, Quadriceps Femoris muscle strength measurement,2 min walking test, fall effectiveness scale,Fall risk self-assessment scale
- Individuals with COPD who are over the age of 65 and have no history of falling: Individuals with COPD who were over the age of 65 and did not have a history of falling were included in this group.
  Interventions: Other: Changed Medical research Council,Mini Mental Test, Quadriceps Femoris muscle strength measurement,2 min walking test, fall effectiveness scale,Fall risk self-assessment scale

INTERVENTIONS:
Other: Changed Medical research Council,Mini Mental Test, Quadriceps Femoris muscle strength measurement,2 min walking test, fall effectiveness scale,Fall risk self-assessment scale — All individuals were given a respiratory function test to evaluate respiratory functions before and after training Modified Medical research Council to evaluate dyspnea, Mini Mental Test to evaluate cognitive status
  , Berg Balance Test to evaluate balance, 2-minute walk test to evaluate walking speed. A hand dynamometer will be used to measure QuadricepsFemoris muscle strength, Fall efficiency scale Fall risk self-assessment scale will be used to evaluate falls.

SUMMARY:
A descriptive study evaluating balance, gait speed, Quadriceps Femoris muscle strength and quality of life in individuals with Chronic obstructive pulmonary disease (COPD) who fell and did not fall.

DETAILED DESCRIPTION:
Falls in the elderly can have devastating consequences. The ability to maintain stability and balance is critical for functional independence, mobility, and avoidance of falls in activities of daily living. An impaired balance is associated with an increased risk of falls and causes a higher mortality rate among older adults. Balance impairment is independently associated with falls in patients with Chronic obstructive pulmonary disease. Well-known risk factors for falls in individuals with Chronic obstructive pulmonary disease include advanced age, increased comorbidities, dyspnea, physical inactivity, muscle weakness, fear and decreased balance confidence, as well as lower extremity muscle weakness. It has been reported that there are functional deficiencies, lack of performance and postural control. According to the results of a recent study, it was found that Chronic obstructive pulmonary disease is in the second place after osteoarthritis in chronic conditions where the prevalence of falls is highest. The prevalence of falls in individuals with Chronic obstructive pulmonary disease is estimated to range from 25% to 46%.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD according to criteria
* Not having had an attack in the last 2 months
* Volunteering to participate in the study
* Being 65 years or older
* Not having any mental or communication problems that prevent filling out the surveys to be used in the research.

Exclusion Criteria:

* Having unstable COPD
* Unstable angina, previous Myocardial Infarction, uncontrolled hypertension, cancer, neurological or musculoskeletal diseases with functional limitations
* Being currently addicted to alcohol or drugs
* Being in the process of COPD exacerbation
* Having severe vision and hearing problems
* Having severe cognitive impairment
* Having had major surgery in the last few months

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals with COPD over the age of 65
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Fall Effectiveness Scale | 15.04.2023-30.09.2024
  It contains 10 questions. Each question is given a score between 1-10. 1 point means very confident, 10 points means not at all confident. A patient with a score above 70 is said to have a fear of falling.

SECONDARY OUTCOMES:
To measure balance Berg Balance Scala | 15.04.2023-30.09.2024
  To assess balance. The highest score is 56, scores between 0-20 indicate that the balance is disrupted, 21-41 indicates that the balance is acceptable, and 41-56 indicates that the balance is good.
Quadriceps Femoris muscle strength falling and non-falling individuals with COPD | 15.04.2023-30.09.2024
  We measure the strength of the muscle by applying pressure from the knee with the help of a hand dynamometer.
Two Minute Walk Test | 15.04.2023-30.09.2024
  The patient walks the longest distance he can in 2 minutes and the value is recorded in meters. The aim is to measure the patient's functional capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirikkale High Specialization Hospital, Kırıkkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No